CLINICAL TRIAL: NCT00462267
Title: Examining the Feasibility of Collaborative Care Treatment for Overweight Adolescents
Acronym: SHINE-Garfield
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Garfield Memorial Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101-9295
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Overweight
Keywords: Nutrition; Exercise; Body mass index; Lifestyle change; Obesity; Overweight; Adolescents; Teens
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Enriched lifestyle intervention (Experimental)
  Interventions: Behavioral: Enriched lifestyle intervention

INTERVENTIONS:
Behavioral: Enriched lifestyle intervention — Multi-component lifestyle intervention
  Arms: Enriched lifestyle intervention

SUMMARY:
This project will examine the effectiveness of a primary care based intervention to help overweight teen girls adopt healthy lifestyle practices. Participants will be adolescent females from Kaiser Permanente Northwest primary care clinics with a body mass index above the 90th percentile. Teens will be randomly assigned to (1) a behavioral weight control program (enriched intervention), (2) brief primary care counseling (low intensity intervention), or (3) usual-care (control). For both of the project's active intervention arms, teens' primary care providers will be given customized plans describing the teen's eating and physical activity habits and instructions on how to best work with these teens and their families. The behavioral weight control program will be specifically tailored for teen girls and will include separate group meetings for teens and parents, follow-up telephone contacts with their group leader, and coordinated feedback from the teen's primary care provider.

DETAILED DESCRIPTION:
Overweight / obesity among youth has recently been declared a "public health crisis" in the United States and other Western countries due to its alarming increase in prevalence (Flegal, 1999; Kohn & Booth, 2003; Lobstein et al., 2004; Sokol, 2000). Over the past decade, overweight in youth (Body mass index [BMI] > 95th percentile) has increased 4% for school-age children, 6 - 11 years old. Adolescents, 12 - 19 years of age are even more overweight (5%) (Ogden et al., 2002). Further, American adolescents had the highest prevalence of overweight among 15 western countries included in a cross-sectional, nationally representative school-based study (Lissau et al., 2004). Such trends are particularly troubling given the psychosocial and physical health risks associated with being overweight in childhood (Must & Strauss, 1999). Overweight among youth appears to confer longer-term health risks even among later normative weight adults (Must et al., 1992). Further, both longer-term health risks and the probability of adult obesity is greater for overweight adolescents than for those developing weight problems earlier in childhood (Must et al., 1992; Whitaker et al., 1997). Collectively, these factors suggest adolescent weight control is an important public health priority.

Clinic-based weight control treatments for youth have demonstrated some success, however, most empirically-supported interventions have been designed for younger school-age children and their families (see Epstein et al., 1998 for a review). Even though a large volume of research explores adult-weight control (see NIH-NHLBI, 1998 for a review) and (though more limited) substantial research examines childhood obesity (see Epstein et al., 1998 for a review), obesity treatments for adolescents have not been adequately studied. Furthermore, almost all empirically tested weight control interventions among youth have been based in academic research clinics rather than the primary care medical settings, in which weight problems among these youth are most often identified and, arguably, in which they could be most efficiently treated. Placing adolescent weight-related interventions within primary medical care settings could make such interventions both more cost-effective and easier to disseminate. The purpose of this study is to assess the feasibility, acceptability, relative cost, and efficacy of a collaborative primary care-based behavioral lifestyle intervention (Enriched Intervention - EI) for overweight adolescent females and their families. This multi-component intervention, adapted for gender and developmental stage, will include a combination of assessment, group teen and parent sessions, individual telephone-based coaching contact, and a distinct collaborative care component with follow-up visits to the youth's primary care provider [PCP]. Further, we will compare the EI to a low intensity intervention [LII] (assessment and information about healthy diet and activity, and follow-up visits with the youth's PCP) and a usual care control condition.

We hypothesize that:

1. Adolescents participating in the Enriched Intervention (EI) will have a greater decrease in BMI percentile scores than adolescents receiving the Low Intensity Intervention (LII) or Usual Care.
2. Adolescent in EI will have improved healthy lifestyle skills (e.g., more physical activity, less junk food and sodas) compared with those receiving LII or Usual Care.
3. Adolescents in EI will report higher psychosocial functioning and quality of life outcomes than those receiving LII or Usual Care.
4. Neither intervention will result in increases in problematic eating or weight-related behaviors or beliefs.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 90th percentile or greater
* One or both parent(s) willing to participate in study assessments and parent sessions

Exclusion Criteria:

* Body mass index 99th percentile or greater
* Significant cognitive impairment
* Current pregnancy
* Congenital heart disease that limits activity
* Serious asthma requiring oral prednisone
* Taking medications that increase appetite

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 2 years

SECONDARY OUTCOMES:
Quality of life (PedsQL 4.0) | 2 years
Self esteem (RSE) | 2 years
Depression (PHQ-A) | 2 years
Unhealthy eating practices (QEWPR-A, TFEQ) | 2 years
Weight and shape concerns (WCS) | 2 years
Sociocultural attitudes toward appearance (SATAQ) | 2 years
Participant satisfaction with the intervention | 2 years
Dietary intake | 2 years
Personal and family eating patterns | 2 years
Physical activity | 2 years
Sedentary behaviors | 2 years
Personal and family physical activity patterns | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lynn L DeBar, PhD, MPH, Principal Investigator — Kaiser Permanente; Michelle H Forest, PhD, Study Director — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States